CLINICAL TRIAL: NCT04000906
Title: A Phase Ib Trial of Intraperitoneal Cisplatin and Nab-paclitaxel Administered by Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) in the Treatment of Advanced Malignancies Confined to the Peritoneal Cavity
Brief Title: PIPAC With Nab-paclitaxel and Cisplatin in Peritoneal Carcinomatosis
Acronym: Nab-PIPAC
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Intidhar Labidi-Galy, MD, PhD, Staff Physician, University Hospital, Geneva
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2018-01327-Nab-PIPAC
Record Dates: First submitted 2019-05-29; First posted 2019-06-27 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Peritoneal Carcinomatosis
Keywords: pancreatic cancer; oeso-gastric cancer; epithelial ovarian cancer; primitive peritoneal mesothelioma
MeSH Terms: conditions — Peritoneal Neoplasms; Pancreatic Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Taxes; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): Pressurized intraperitoneal aerosol chemotherapy (PIPAC) administration of Nab paclitaxel and cisplatin
  Interventions: Drug: Nab paclitaxel; Drug: Cisplatin

INTERVENTIONS:
Drug: Nab paclitaxel — Dose escalation (7.5 mg/m2, 15 mg/m2, 25 mg/m2, 37.5 mg/m2, 52.5 mg/m2 and 70 mg/m2)
Drug: Cisplatin — 10.5 mg/m2

SUMMARY:
Phase Ib trial including investigating the combination of nab-paclitaxel and cisplatin in patients diagnosed with peritoneal carcinomatosis related to pancreatic, oeso-gastric, ovarian cancer or primitive peritoneal mesothelioma.

DETAILED DESCRIPTION:
Phase Ib trial investigating the combination of intraperitoneal Cisplatin (10.5 mg/m2) and Nab-paclitaxel (escalated dose from 7.5 mg/m2 to 70 mg/m2) administered by pressurized intraperitoneal aerosol chemotherapy (PIPAC) every 4-6 weeks for 3 cycles.

ELIGIBILITY:
Inclusion criteria:

* Informed consent as documented by signature
* ≥18 years,
* psychologically able to follow the trial procedures
* with peritoneal carcinomatosis from pancreatic, oesogastric, epithelial ovarian cancers or primitive peritoneal mesothelioma,
* ECOG 0, 1 or 2,
* Life expectancy > 3 months,
* Not candidate for surgical cytoreduction and IP/HIPEC based on expert multidisciplinary board
* who received at least one line of chemotherapy and for whom standard therapies have been exhausted or not feasible. patients with residual disease following the first line of therapy or Following secondary debulking are eligible.

Exclusion criteria:

* Predominant extra-peritoneal metastases at the discretion of the study team after discussion at the multidisciplinary board,
* Bowel obstruction, active gastro-duodenal ulcer or ongoing abdominal infection (bacterial, viral or fungal),
* Chemotherapy or surgery within the last two weeks prior to enrollment,
* Previous intra-abdominal chemotherapy,
* General or local (abdominal) contra-indications for laparoscopic surgery
* Known allergy to cisplatin or other platinum-containing compounds or to nab-paclitaxel,
* Severe renal impairment (calculated GFR (CKD-EPI) < 60 mL/min/1.73 m2), myelosuppression (platelet count < 100.000/μl, hemoglobin < 9g/dl, neutrophil granulocytes < 1.500/ml), International Normalized Ratio (INR) > 2, severe hepatic (Serum total bilirubin > 1.5 mg/dl), respiratory or neurologic impairment (grade 3), severe myocardial insufficiency (NYHA class > 2), recent myocardial infarction, severe arrhythmias,
* Pregnancy or breastfeeding, women who can become pregnant must ensure effective contraception.
* Known or suspected non-compliance, inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Determine the maximal tolerated dose (MTD) of Nab paclitaxel (Abraxane®) administered IP by PIPAC in concomitance with cisplatin. | From the time of treatment randomization through 30 days following cessation of treatment
  MTD is defined as the lowest dose level at which ≥33% of patients' experience dose limiting toxicity in accordance to CTCAE version 5.0 criteria.

SECONDARY OUTCOMES:
Adverse events (AE) and serious adverse events (SAE) | D-1/D10 of each cycle
  AE and SAE with predefined toxicity criteria will be applied using CTCAE version 5.0 criteria, documented before and after each cycle of PIPAC treatment. Surgical complications will be assessed according to Clavien classification and comprehensive complication index (CCI)
The efficacy | D0 of each cycle
  It will be assessed by the objective histological regression and objective tumor response rate (OTR) according to the new regression system for peritoneal cancer (PRGS, peritoneal regression grade score system). The objective response rate (ORR), the clinical benefit rate (CBR) as defined by RECIST version 1.1 criteria and the relevance of radiological response assessed by CT enterography (CT-PCI score).
The QoL | D-1/D10 of each cycle
  QoL will be evaluated based on the EORTC questionnaire QLQ-C30 Version 3.0 and visual analogic scale for pain (VAS scale).

CONTACTS AND LOCATIONS:
Overall Officials: Intidhar Labidi-Galy, MD, PhD, Principal Investigator — University Hospital, Geneva
Locations (2):
- Switzerland (2):
  - University Hospital, Lausanne, Lausanne, Canton of Vaud
  - University Hospital, Geneva, Geneva

IPD SHARING:
Plan to Share IPD: Yes
The only clinical data available to researchers will be anonymised. Requests may be directed to Sponsor Investigator or designee. The informed consent form and clinical study report will be made available
Supporting Information: ICF, CSR
Time Frame: Data can be shared no earlier than 1 year following the date of publication.
Access Criteria: All data supporting the findings of the current study will be made available from the corresponding author upon reasonable request.

REFERENCES:
- [Derived] Lang N, Diciola A, Labidi-Galy I, Ris F, Di Marco M, Mach N, Petignat P, Toso C, Undurraga M, Hubner M. Nab-PIPAC: a phase IB study protocol of intraperitoneal cisplatin and nab-paclitaxel administered by pressurised intraperitoneal aerosol chemotherapy (PIPAC) in the treatment of advanced malignancies confined to the peritoneal cavity. BMJ Open. 2023 Jan 5;13(1):e067691. doi: 10.1136/bmjopen-2022-067691. PMID 36604127